CLINICAL TRIAL: NCT01142479
Title: The Effects of Compound Herbal Formula(TPE-1) for Leukopenia and Cancer-related Fatigue in Breast Cancer Patients With Radiotherapy
Brief Title: Compound Herbal Formula (TPE-1) for Leukopenia and Cancer-related Fatigue in Breast Cancer Patients With Radiotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chung-Hua Hsu, vice superintendent, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPE-1-breast Ca
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer; Radiotherapy; Chinese Herbal Medicine
Keywords: Breast Cancer; Radiotherapy; Chinese herbal medicine; TPE-1; Leukopenia
MeSH Terms: conditions — Breast Neoplasms; Leukopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- herbal A (Placebo Comparator): dilute of (TPE-1) decoction.
  Interventions: Drug: Chinese herbal medicine decoction
- herbal B (Experimental): TPE-1 decoction (100 ml)
  Interventions: Drug: Chinese herbal medicine decoction

INTERVENTIONS:
Drug: Chinese herbal medicine decoction — 100 ml /Qd for 6 weeks(42 days)
  Other Names: TPE-1

SUMMARY:
Many breast cancer patients will taking Chinese herbal medicine during receiving radiotherapy. The investigators conducted the pilot study showing Compound Herbal Formula (TPE-1) have the effect of improving the fatigue and leukopenia during radiotherapy. So the investigators designed this double blind and controlled trial to evaluate whether TPE-1 have the effects for leukopenia and cancer-related fatigue in breast cancer patients with radiotherapy. From our initial observation for 2 years, TPE-1 is safety. The study is also designed to evaluate the safety when patients taking this formula.

DETAILED DESCRIPTION:
TPE-1 is designed according to TCM concept. It is not anti-cancer directly, it is enhancing the Qi flow and immunity of breast cancer when they are just finishing chemotherapy and on going radiotherapy. Many Chinese population will seeking Chinese herbal medicine under the same condition.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* age between 18 to 70 yrs
* finished chemotherapy (adriamycin ), will receiving radiotherapy
* Chinese population
* KP$ between 40-100
* ECOG < 2
* WBC >4X10(9)／L and Hb > 10g/dl
* Assigned informed concent.

Exclusion Criteria:

* receiving operation during 14 days
* blood transfusion during one month.
* ALT >100mg/dL
* Creatinine >2.0mg/dL
* Total bilirubin >2.0mg/dL
* Infection
* prolation
* Taking anti-seizure , psychological drugs or any drugs not suitable patients
* AIDS or any disease diagnosed by physician and not suitable patients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
the % change of white blood cell(WBC) count | 6 weeks
  WBC will be checked before taking TPE ans after taking TPE-1.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | 6 weeks
  The Hb will be checked before and after kaking TPE-1

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, Taipei, Taiwan, Taiwan